CLINICAL TRIAL: NCT00825123
Title: The Influence of Heart Rate Reduction Upon Central Arterial Pressure in Younger and Older Healthy Individuals
Brief Title: Effects of Heart Rate Reduction on Central Arterial Pressure in Healthy Individuals
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 141/07 bayside health
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2009-11

CONDITIONS: Central Arterial Pressure
Keywords: healthy individuals
MeSH Terms: interventions — Ivabradine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ivabradine (Experimental)
  Interventions: Drug: Ivabradine
- Metoprolol (Active Comparator)
  Interventions: Drug: Metoprolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 10 mg once
  Other Names: Coralan
  Arms: Ivabradine
Drug: Metoprolol — Metoprolol 50 mg once
  Arms: Metoprolol
Drug: Placebo — Lactose powder
  Arms: Placebo

SUMMARY:
The purpose of this project is to determine the effects of slowing heart rate upon both central and peripheral blood pressures using Ivabradine. The effects of Ivabradine will be compared to Metoprolol and placebo.

Participants will attend the hospital for 3 visits where they will be randomised to receive either Ivabradine, Metoprolol and placebo on each visit. Non-invasive measures of blood pressure will be recorded before and after consuming the study drug.

DETAILED DESCRIPTION:
Participants will undergo three days of laboratory testing, each visit separated by at least seven days.

In order to assess each potential participant's suitability for the study based upon the relevant inclusion and exclusion criteria, the first visit will involve a medical consultation (history and physical examination), venepuncture (for full blood examination, lipid profile and biochemistry) and a 12-lead surface electrocardiogram. Baseline measurements of central and peripheral arterial and pulse wave velocity will be made at baseline, and 4 hours following the administration of either placebo, 50mg of metoprolol or a 10mg oral dose of ivabradine. The placebo will contain lactose powder.

Subjects will be randomized according to a 3-by-3 Latin square design. Central pulse pressure will be assessed using carotid artery tonometry using a non-invasive Millar Mikro-tip pressure transducer. The transducer is used to applanate the carotid artery and calibrated using brachial mean and diastolic blood pressure (automated oscillometric sphygmomanometer).

Pressure waveforms will also be recorded at the radial, brachial and femoral arteries to permit study of wave reflection at these sites.

Measurements will be taken be taken before and 4 hours following the oral administration of metoprolol/ivabradine/placebo.

Bias will be minimized by blinding both the participants and research staff responsible for data collection to the administered drug.

Any potential patient-specific confounding factors will have minimal impact, as the same participants will be studied after the administration of the three agents.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* aged 18 - 25 years OR
* aged >60 years

Exclusion Criteria:

* Chronic disease
* Unable to give informed consent
* Treated or untreated systemic arterial hypertension (SBP >160mmHg and/or DBP > 90mmHg)
* Resting bradycardia (heart rate < 60 beats/minute)
* Pregnancy or active lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11-08 (Actual); Study Completion 2011-11-08 (Actual)

PRIMARY OUTCOMES:
central arterial pressure | baseline and 4 hours post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker IDI Hearte & Diabetes Institute
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia